CLINICAL TRIAL: NCT00583063
Title: A Pharmacokinetic Interaction Study of Rapamycin (Sirolimus) and SU11248 (Sunitinib) in Patients With Advanced Solid Tumors
Brief Title: Interaction Study of Rapamycin and Sunitinib in Patients With Advanced Cancers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15328B
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2011-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Sunitinib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Sunitinib taken by mouth every day. Rapamycin (taken by mouth) will be started on Day 15 and then taken every day. Drugs can be taken until disease progression.
  Interventions: Drug: sunitinib; Drug: rapamycin
- B (Experimental): Rapamycin taken by mouth every day. Sunitinib (taken by mouth) will be started on Day 15 and then taken every day. Drugs can be taken until disease progression.
  Interventions: Drug: sunitinib; Drug: rapamycin

INTERVENTIONS:
Drug: sunitinib — 25 mg daily (oral dosing)
  Other Names: Sutent
Drug: rapamycin — 4 mg daily (oral dosing)
  Other Names: Rapamune

SUMMARY:
Determine the pharmacokinetic interactions between rapamycin and sunitinib in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable cancer for which standard treatments do not exist or are no longer effective or cancers where evidence of efficacy of single agent sunitinib or single agent mTOR inhibitor has been demonstrated
* Measurable or non-measurable disease.
* No prior treatments for 4 weeks before starting study
* No ongoing toxicities from previous treatments
* 18 years or older
* Performance status 2 or better
* Life expectancy of at least 3 months.
* Normal organ and marrow function as defined below:

  * No transfusions of packed red blood cells within 1 week of starting treatment. A hemoglobin of 9.0 g/dL or greater is recommended. Patients should not be transfused for protocol participation.
  * Leukocytes greater than or equal to 3,000/μL
  * Absolute neutrophil count greater than or equal to 1,500/μL
  * Platelets greater than or equal to 100,000/μL
  * Total bilirubin less than or equal to 1.5 x ULN
  * AST and ALT less than or equal to 2.5x ULN (less than or equal to 5x ULN if liver function abnormalities are due to underlying disease)
  * Creatinine within normal institutional limits OR
  * Creatinine clearance > 60 mL/min/1.73 m2
  * PT or INR within normal institutional limits
  * Serum calcium within normal institutional limits
* QTc < 500 msec.
* Patients with prior anthracycline exposure or that have received central thoracic radiation must have NYHA class I cardiac function
* Must agree to use adequate birth control
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatments within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of entering the study or those who have not recovered from adverse events due prior treatments
* Current treatment with other investigational agents.
* Prior therapy with a VEGFR or mTOR inhibitor
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rapamycin or sunitinib.
* QTc prolongation (QTc interval equal to or greater than 500 msec) or other significant ECG abnormalities
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture.
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment.
  * Known active infection
  * Major surgery or radiation therapy within 4 weeks of starting the study treatment.
  * NCI CTCAE Version 3.0 grade 3 hemorrhage within 4 weeks of starting the study treatment.
  * History of CVA or transient ischemic attack within 12 months prior to study entry.
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry.
  * History of pulmonary embolism within the past 12 months.
  * Class III or IV heart failure as defined by the NYHA functional classification system
  * Ongoing cardiac dysrhythmias
  * Poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher)
  * Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
  * History of interstitial lung disease
* Patients with severe immunodeficient states (as judged by the treating physician)
* Pregnancy or breastfeeding.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for interactions with the study drugs
* Use of certain medications (as determined by the investigator)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk or interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic interactions | 4 weeks

SECONDARY OUTCOMES:
Toxicity of the combined drug regimen | 4 weeks
Response to drug regimen | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States